CLINICAL TRIAL: NCT03390413
Title: Robot-assisted Surgical Resection vs. Cryoablation of Localised Renal Cancer - a Randomised Trial of Functional, Oncological and Financial Aspects
Brief Title: Robot-assisted Surgical Resection vs. Cryoablation of Localised Renal Cancer
Acronym: ROAST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics and lack of funding
Sponsor: Jørgen Bjerggaard Jensen (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, MD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFE-1-10-72-140-17
Record Dates: First submitted 2017-12-20; First posted 2018-01-04 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Renal Cancer
Keywords: Cryoablation; Robot-assisted surgical resection
MeSH Terms: conditions — Kidney Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robot (Active Comparator)
  Interventions: Procedure: Robot
- Cryo (Experimental)
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Robot — Renal cancer treated with robotic surgery
  Arms: Robot
Procedure: Cryoablation — Renal cancer treated with cryoablation
  Arms: Cryo

SUMMARY:
The present study is a randomized clinical trial which investigates robot-assisted partial nephrectomy (RPN) compared to image-guided cryoablation (CA) in a number of functional, oncological and economic variables.

Every year close to 1000 Danes are diagnosed with renal cell carcinoma. Approximately 25% of these newly diagnosed patients have a T1a tumour, thus being candidates to nephron-sparing surgery. Today most nephronsparing surgical procedures consists of RPN, often requiring temporary clamping of the renal artery rendering the kidney to a critical period of warm ischemia which is potentially harmful to the renal function. Image guided ablative modalities has emerged as a minimal-invasive alternative to partial nephrectomy. The level of evidence within this domain is considered to be low as the existing literature is highly influenced by selection bias, and as of yet no randomized trial has compared the two modalities. Especially with the increasing age of the patients, an approach suitable for local anaestesia is desirable.

Patients from Central Denmark Region and Region of Southern Denmark who are diagnosed with a pT1a renal cell carcinoma that is found to be eligible for both modalities will be offered to enter into a randomized trial to be treated with either RPN og CA. The study's primary endpoint is loss of renal function 6 and 12 month after treatment. Secondary endpoint includes recurrence free survival 1, 3 and 5 years after treatment, readmission and complication rates as well as health economic evaluations.

All patients will be pre- and postoperatively assessed with biochemistry, CT urography, CT thorax and glomerular filtration rate measurements.

DETAILED DESCRIPTION:
The diagnosis and management of renal cell carcinoma (RCC) have changed remarkably rapidly. Although the incidence of RCC has been increasing, survival has improved substantially. As incidental diagnosis of small indolent cancers has become more frequent, active surveillance, robot-assisted nephron-sparing surgical techniques and minimally invasive procedures, such as thermal ablation, have gained popularity. Despite progression in cancer control and survival, locally advanced disease and distant metastases are still diagnosed in a notable proportion of patients.

In 2013, RCC was diagnosed in more than 350.000 people worldwide, making it the seventh most common tumour, and this cancer is associated with more than 140.000 deaths per year. Incidence of RCC varies worldwide, being higher in developed countries than in developing countries. In Europe, mortality from RCC peaked at 4.8 per 100.000 in 1990-94 and had declined to 4.1 per 100.000 (-13%) in 2000-04. In the US, 5-year relative survival rates increased from 50% in 1975-77 to 73% in 2003-09. According to the Danish Cancer Registry, approx. 1000 Danes are annually diagnosed with RCC, of which approx. 25% have a small localised tumour that are potentially eligible for a minimal invasive nephron-sparing treatment modality.

With the expansion of routine imaging for many disorders, patients with RCC are increasingly being identified by chance. Only 30% of patients are diagnosed on the basis of symptoms. Small renal masses (SRM) refers to tumours less than 4 cm I diameter, which have not spread beyond the kidney (T1a tumours). The highest incidence of SRM is seen in patients older than 65 years, who generally present themselves with varying degrees of comorbidity. Thus, minimally invasive treatment modalities are highly relevant in the treatment of RCC in the ever-growing elderly population.

Notwithstanding the advances in the understanding of RCC biology, surgery remains the mainstay of curative treatment. Although radical nephrectomy was the standard of care for the management of renal tumours, the detection of SRMs and accumulating evidence that surgical induced chronic kidney disease can increase patients' morbidity have led to more conservative approaches. Specifically, nephron-sparing surgery, ablative modalities and active surveillance. When treating patients with SRM three competing factors must be considered; comorbidity, renal function and oncological outcome. Active surveillance remains controversial as absolute cut-offs for tumour size and growth rate that should prompt intervention are not well defined. In comparison to radical nephrectomy, nephron-sparing surgery has increasingly been used since observations suggested oncological control similar to radical nephrectomy but with the additional benefit of renal preservation and a reduced risk of cardiovascular events. These functional outcomes become important because patients with organ-confined RCC that has been surgical treated are usually long-term survivors (10-years cancer-specific survival of 85-96%). Today most nephron-sparing surgical procedures consists of robot-assisted partial nephrectomy (RPN).

Although surgery still represents the standard of care for RCC, the use of minimally invasive ablative techniques to treat SRMs has been increasing. Ablative treatment such as cryoablation (CA) were initially contemplated only to patients with a single kidney or those deemed unfit to more extensive surgical procedures. Since an increasing number of reports have shown acceptable oncological control and low complications rates the clinical indications for these procedures has been extending. Most studies of outcomes after CA consist of single-institution retrospective reports with low number of un-randomised patients with short follow-up.

Compared to RPN the ablative modalities offer several advantages. Most ablative procedure are now performed as an image-guided procedure on an outpatient basis without the need for surgical intervention. Furthermore, many RPN-procedures requires temporary clamping of the renal artery which renders the kidney to a critical period of warm ischemia.

There exist only very few reports comparing surgical modalities to ablative modalities but a systematic review and meta-analysis of six clinical trials showed that recurrence-free survival and cancer-specific survival were similar for patients treated with surgery or ablation, with less postoperative decline in estimated glomerular filtration rate in the ablation group. The overall complication rate was significantly lower in the ablation group. The existing literature are highly influenced by selection bias and ss of yet no randomised trial has compared RPN to CA.

Since 2015 the treatment of RCC has been located at two centers in Region Midtjylland, Hospitalsenheden Vest Holstebro were RPN are being performed and Aarhus University Hospital were CA are being performed. Both treatment modalities are considered highly expensive with financial costs in the area of dkr. 30.000 to 50.000.

ELIGIBILITY:
Inclusion Criteria:

* First-time biopsy confirmed RCC
* ECOG Performance Status between 0 and 2
* The tumour is found to be eligible for both RPN and CA
* e-GFR> 60 ml/min/1.74 m2
* Written consent after oral and written information has been given

Exclusion Criteria:

* Impaired renal function (e-GFR <59 ml/min/1.74m2)
* Previously diagnosed with RCC
* Patients with recognized genetic mutations that directly relate to RCC (eg. Von Hippel Lindau, BHD)
* Allergy to contrast agents
* Pregnancy
* Expected remaining life <12 months
* Active treatment of secondary cancer disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Renal function | 6 months
  Loss of renal function measured by Chrome-EDTA clearence 6 months post-operatively in each treatment modality

SECONDARY OUTCOMES:
Incomplete ablation | 3 months
  The degree of incomplete ablation 3 months after CA in comparison with the degree of positive surgical margin by robot-assisted resection
Complications | 90 days
  Number of treatment related complications up to 90 days after treatment
Costs | 90 days
  Treatment related costs evaluated by micro costing

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitropoulos D, Artibani W, Biyani CS, Bjerggaard Jensen J, Roupret M, Truss M. Validation of the Clavien-Dindo Grading System in Urology by the European Association of Urology Guidelines Ad Hoc Panel. Eur Urol Focus. 2018 Jul;4(4):608-613. doi: 10.1016/j.euf.2017.02.014. Epub 2017 Mar 7. PMID 28753862
- [Background] Vind-Kezunovic S, Bouchelouche K, Ipsen P, Hoyer S, Bell C, Bjerggaard Jensen J. Detection of Lymph Node Metastasis in Patients with Bladder Cancer using Maximum Standardised Uptake Value and 18F-fluorodeoxyglucose Positron Emission Tomography/Computed Tomography: Results from a High-volume Centre Including Long-term Follow-up. Eur Urol Focus. 2019 Jan;5(1):90-96. doi: 10.1016/j.euf.2017.06.005. Epub 2017 Jun 23. PMID 28753817
- [Background] Nielsen TK, Jensen JB. Efficacy of commercialised extracorporeal shock wave lithotripsy service: a review of 589 renal stones. BMC Urol. 2017 Jul 27;17(1):59. doi: 10.1186/s12894-017-0249-8. PMID 28750620